CLINICAL TRIAL: NCT06979427
Title: Evaluation of the Ability of CTFFR to Determine Non-significant Lesions of Coronary Disease Based on MACE in One-year Follow-up of Patients (Seeing Beyond the Stenosis: CTFFR and MACE in a One-Year Follow-Up)
Brief Title: CTFFR and Prediction of Non-Significant CAD Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Kojuri, professor, Shiraz University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 1403.414
Record Dates: First submitted 2025-05-16; First posted 2025-05-19 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Chronic Coronary Syndrome
Keywords: Chronic Coronary Syndrome; Major adverse coronary events (MACE); fractional flow reserve; coronary CT angiography

STUDY DESIGN:
Intervention Model Description: NIFFR of coronary less than 0.8
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nonsignificant NIFFR (Experimental): patients with coronary artery lesion in CT angiography, with NIFFR of more than 0.8
  Interventions: Diagnostic Test: NIFFR
- significant NIFFR (Active Comparator): patients with coronary artery lesion in CT angiography, with NIFFR of more than 0.8
  Interventions: Diagnostic Test: NIFFR

INTERVENTIONS:
Diagnostic Test: NIFFR — Fractional flow reserve derived from CT angiography from lesion between 50-70%
  Other Names: Non invasive fractional flow reserve

SUMMARY:
In this prospective cohort study, 250 patients with suspected or known CAD and at least one intermediate coronary lesion (50-70% stenosis) who had a NiFFR value greater than 0.80 underwent coronary computed tomography angiography (CCTA) with NiFFR assessment. Patients were followed for one year to monitor for MACE

DETAILED DESCRIPTION:
This prospective cohort includes people with known or suspected CAD who had both CCTA and ICA with this index (FFR) measurements. Patients were enrolled if they had at least one intermediate coronary lesion (classified as 50-70% diameter stenosis on visual judgment) on CCTA and then underwent FFR testing.

Data about the patients was acquired from the Professor Kojuri registry. The database provided demographic information for instance age, gender, CAD family history, prior CAD history, hypertension (HTN), diabetes mellitus (DM), and hyperlipidaemia (HLP). The prevalence of cigarette smoking and the ejection fraction of the left ventricle. Lesion and Vessel Characteristics were also collected from registry.

The target vessel was identified (LAD, RCA, LCX, or LMC), the lesion was located (proximal, mid, or bifurcation), the vessel diameters were measured (proximal, distal, stenotic), and the lesion length was determined. Measurements were taken using CCTA datasets using semi-automated software methods.

Patients were clinically monitored for one year after examination. The primary outcome was the occurrence of major cardiovascular consequences, or MACE, which included cardiac-related death, acute coronary syndrome (ACS), unexpected revascularisation, and hospitalization for cardiac reasons. Throughout the one-year study period, all participants were visited every three months and followed up with phone calls.

ELIGIBILITY:
Inclusion Criteria:

* Patients were enrolled if they had at least one intermediate coronary lesion (classified as 50-70% diameter stenosis on visual judgment) on CCTA and then underwent FFR testing

Exclusion Criteria:

* Patients having past coronary artery bypass graft surgery (CABG)
* previous PCI in the target vascular
* significant renal impairment define with eGFR < 30 mL/min/1.73 m²
* contrast allergy
* poor image quality that prevented appropriate CCTA or CT-FFR analysis

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with MACE | 1 year
  Number of patients with Major adverse cardiac events,which included cardiac-related death, acute coronary syndrome (ACS), unexpected revascularisation, and hospitalization for cardiac reasons, stroke
Number of patients with bleeding | 1 year
  Number of patients with major or minor bleeding based on BARC classification

SECONDARY OUTCOMES:
Number of patients with dyspnoea | 1 year
  Number of patients with minor and major dyspnoea ( based on that it affect daily activity or tolerable or not)

CONTACTS AND LOCATIONS:
Locations (1):
- Professor Kojuri Cardiology Clinic, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: No
data sharing by rational request